CLINICAL TRIAL: NCT01288235
Title: A Phase II Study of Proton Radiotherapy for Pediatric Brain Tumors Requiring Partial Brain Irradiation: An Assessment of Long Term Neurocognitive, Neuroendocrine Adn Ototoxicity Outcomes
Brief Title: Proton Radiotherapy for Pediatric Brain Tumors Requiring Partial Brain Irradiation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Torunn Yock, MD, Director, Pediatric Radiation Oncology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-206
Record Dates: First submitted 2011-02-01; First posted 2011-02-02 (Estimated); Results first posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Brain Tumor; Low Grade Glioma; Astrocytoma; Ependymoma; Ganglioglioma
Keywords: proton radiotherapy
MeSH Terms: conditions — Brain Neoplasms; Astrocytoma; Ependymoma; Ganglioglioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Proton Radiotherapy (Experimental): Proton Radiotherapy
  Interventions: Radiation: Proton radiotherapy

INTERVENTIONS:
Radiation: Proton radiotherapy — 5 days a week

SUMMARY:
Some patients with brain tumors receive standard radiation to help prevent tumor growth. Although standard radiation kills tumor cells, it can also damage normal tissue in the process and lead to more side effects. This research study is looking at a different form of radiation called proton radiotherapy which helps spare normal tissues while delivering radiation to the tumor or tumor bed. Proton techniques irradiate 2-3 times less normal tissue then standard radiation. This therapy has been used in treatment of other cancers and information from those other research studies suggests that this therapy may help better target brain tumors then standard radiation.

DETAILED DESCRIPTION:
- Participants will receive proton radiotherapy at the Francis H. Burr Proton Therapy Center which is located at the Massachusetts General Hospital. They will receive the proton radiotherapy 5 days per week. The number of weeks the participant will be receiving proton radiotherapy depends upon the tumor type and location and how well they are tolerating the treatment. Participant's will have a physical exam weekly during proton radiotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven low grade glioma or astrocytoma, ependymoma, craniopharyngioma, meningioma, neurocytoma, medulloblastoma or gangliogliomas or other rare tumor requiring tumor bed or tumor irradiation. Patients with a presumed diagnosis of optic glioma or gliomas based on imaging and clinical characteristics will also be allowed on this trial.
* Patients with biopsy proven high grade glioma (excluding GBM) and a gross total resection and patients with non-disseminated atypical teratoid rhabdoid (ATRT) may also be included.
* Pathologic diagnosis must be based on pathology or pathology review by Department of Pathology at MGH or another DF/HCC institution.
* Age between 1-25 years.
* Life expectancy of greater than 1 year.
* ECOG Performance Status 0, 1, 2 or 3 or Lansky performance status 30 or greater.
* Girls and women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.

Exclusion Criteria:

* Participants who have had radiotherapy to the site to be treated.
* Participants with known spinal or distant metastases. Patients with ependymoma, medulloblastoma or germinoma must have metastatic workup including spine MRI to rule out metastases.
* Uncontrolled intercurrent illness that would limit compliance with study requirements.
* Pregnant or breastfeeding women.
* Patients who cannot participate in contributing to the neurocognitive outcomes due to severe neurologic impairment or language barrier (ie not English or Spanish speaking) will be excluded from this study.

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Torunn I. Yock, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Vatner RE, Niemierko A, Misra M, Weyman EA, Goebel CP, Ebb DH, Jones RM, Huang MS, Mahajan A, Grosshans DR, Paulino AC, Stanley T, MacDonald SM, Tarbell NJ, Yock TI. Endocrine Deficiency As a Function of Radiation Dose to the Hypothalamus and Pituitary in Pediatric and Young Adult Patients With Brain Tumors. J Clin Oncol. 2018 Oct 1;36(28):2854-2862. doi: 10.1200/JCO.2018.78.1492. Epub 2018 Aug 17. PMID 30118397

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Proton Radiotherapy
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Proton Radiotherapy
Number analyzed (Participants) | 100
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 8.0 [3.5 to 13.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 80
  More than one race | 4
  Unknown or Not Reported | 13
Region of Enrollment [Number; unit: participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: Endocrine Dysfunction
Description: Cumulative incidence (estimated percentage participants) that developed endocrine dysfunction at 3- and 5-years following completion of proton radiation therapy.
Time Frame: 3- and 5- years post radiation treatment
Population: Patient population at risk of developing an endocrine dysfunction during follow-up
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Proton Radiotherapy
Number analyzed (Participants) | 99
percentage of participants
  3-Years post RT | 14.5 [8.3 to 22.3]
  5-Years post RT | 20.2 [12.7 to 28.9]
Statistical Analysis 1: Comparison: Proton Radiotherapy; Test type: Other; 3-Year Cumulative incidence = 14.5, 95% CI 2-sided [8.3 to 22.3]
Statistical Analysis 2: Comparison: Proton Radiotherapy; Test type: Other; 5-Year Cumulative incidence = 20.2, 95% CI 2-sided [12.7 to 28.9]

2. Primary Outcome: Neurocognitive Sequelae
Description: The overall change in neurocognitive outcomes between treatment and last-follow-up as assessed by Wechsler Intelligence Scale for Children version 4 (WISC-IV). The test measures the Full-Scale Intelligence Quotient (FSIQ) of children through four indices; the Verbal Comprehension Index (VCI), Perceptual Reasoning Index (PRI), working memory test, and a processing speed test. FSIQ and the four indices are all assessed on a bell curve scale with an average score of 100 and standard deviation of 15. Higher scores represent higher intelligence and lower scores represent reduced intelligence.
Time Frame: From the start of radiation treatment (baseline) to study completion. Participants were assessed annually up to 5 years following treatment completion. The median follow-up is 4.7 years.
Population: Patients who received neurocognitive testing at both baseline and post radiation treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Proton Radiotherapy
Number analyzed (Participants) | 49
score on a scale
  Baseline FSIQ | 99.2 (14.8)
  Latest Follow-up FSIQ | 100.3 (16.2)
Statistical Analysis 1: Comparison: Proton Radiotherapy; Test type: Other; p = 0.543, t-test, 2 sided; Paired t test; Mean Difference (Net) = 1.1, 95% CI 2-sided [-2.6 to 4.9]

3. Secondary Outcome: Disease Control
Description: Three and 5 year local and distant disease control survival probabilities. Participants were assessed each follow-up and categorized in the following ways: 1) disease controlled no evidence of progression, 2) disease not controlled, tumor has progressed 3) patient has suffered a second malignancy (new tumor unrelated to the one the participant was treated for). Disease failure (recurrence of primary tumor) can occur locally (at or near the site of the original tumor), distally (located further away from the original tumor site), or both.
  Participants who did not fail locally or in a distant site were censored at the date of their last follow-up, including death due to other causes. Disease control shows the percent probability of remaining recurrence free (disease is controlled) in follow-up post radiation treatment completion.
Time Frame: 3- and 5- years post radiation treatment
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Proton Radiotherapy
Number analyzed (Participants) | 100
percent probability
  Local Control 3-Year post RT | 89.9 [83.1 to 94.9]
  Local Control 5-Year post RT | 85.9 [78.2 to 91.9]
  Distant Control 3-Year post RT | 97.0 [92.1 to 99.2]
  Distant Control 5-Year post RT | 95.0 [89.4 to 98.1]
Statistical Analysis 1: Comparison: Proton Radiotherapy; Test type: Other; 3-Year Local Disease Control Probability = 89.9, 95% CI 2-sided [83.1 to 94.9]
Statistical Analysis 2: Comparison: Proton Radiotherapy; Test type: Other; 5-Year Local Disease Control Probability = 85.9, 95% CI 2-sided [78.2 to 91.9]
Statistical Analysis 3: Comparison: Proton Radiotherapy; Test type: Other; 3-Year Distant Disease Control = 97.0, 95% CI 2-sided [92.1 to 99.2]
Statistical Analysis 4: Comparison: Proton Radiotherapy; Test type: Other; 5-Year Distant Disease Control = 95.0, 95% CI 2-sided [89.4 to 98.1]

4. Secondary Outcome: Cumulative Incidence of Grade 3+ Toxicities
Description: Percentage of participants who experienced a toxicity following completion of radiation treatment as measured by the NCI Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE 4.0) after the completion of radiation therapy. Cumulative incidence is shown at 3- and 5-years post treatment. The descriptions and grading scales found in the NCI Common Terminology Criteria
Time Frame: 3- and 5- years post radiation treatment
Population: Patients at risk of developing a grade 3 or higher toxicity following proton radiation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Proton Radiotherapy
Number analyzed (Participants) | 99
percentage of participants
  3-Years post RT | 12.2 [6.6 to 19.5]
  5-Years post RT | 16.3 [9.8 to 24.3]
Statistical Analysis 1: Comparison: Proton Radiotherapy; Test type: Other; 3-Year Cumulative incidence of grade 3+ = 12.2, 95% CI 2-sided [6.6 to 19.5]
Statistical Analysis 2: Comparison: Proton Radiotherapy; Test type: Other; 5-Year Cumulative incidence of grade 3+ = 16.3, 95% CI 2-sided [9.8 to 24.3]

5. Secondary Outcome: Cumulative Incidence of Ototoxicity
Description: Cumulative incidence (estimated percentage participants) who experienced ototoxicity defined as either grade 3 or 4 hearing loss in either ear after the completion of radiation therapy in the overall participant population. Cumulative incidence and 95% confidence intervals are shown at 3- and 5-years post radiation treatment.
Time Frame: 3- and 5- years post radiation treatment
Population: Patients with audiograms completed at both baseline and follow-up and at risk of developing grade 3 or 4 high grade hearing loss in either ear after radiation treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Proton Radiotherapy
Number analyzed (Participants) | 28
percentage of participants
  3-Years post RT | 12.5 [2.9 to 29.5]
  5-Years post RT | 12.5 [2.9 to 29.5]
Statistical Analysis 1: Comparison: Proton Radiotherapy; Test type: Other; 3-Year Cumulative inc. of hearing loss = 12.5, 95% CI 2-sided [2.9 to 29.5]
Statistical Analysis 2: Comparison: Proton Radiotherapy; Test type: Other; 5-Year Cumulative inc. of hearing loss = 12.5, 95% CI 2-sided [2.9 to 29.5]

ADVERSE EVENTS:
Time Frame: All adverse events, both serious and non-serious, and deaths were collected from the initiation of study intervention, during treatment, and annually for up to 5 years after the completion of radiation treatment.
Description: Toxicity assessments were done using NCI Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Arm/Group | Proton Radiotherapy
All-Cause Mortality (participants affected / at risk) | 15/100
Serious Adverse Events (participants affected / at risk) | 2/100
Other Adverse Events (participants affected / at risk) | 98/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Proton Radiotherapy (N=100)
Hypernatremia (Metabolism and nutrition disorders) | 1
Lymphocyte Count Decreased (Investigations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Proton Radiotherapy (N=100)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 3
Ear pain (Ear and labyrinth disorders) | 2
External ear pain (Ear and labyrinth disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 8
Middle ear inflammation (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 8
Delayed puberty (Endocrine disorders) | 1
Endocrine disorders - Other (Endocrine disorders) | 22
Hyperthyroidism (Endocrine disorders) | 1
Hypoparathyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 8
Precocious puberty (Endocrine disorders) | 4
Blurred vision (Eye disorders) | 4
Cataract (Eye disorders) | 1
Eye disorders - Other (Eye disorders) | 14
Eyelid function disorder (Eye disorders) | 1
Optic nerve disorder (Eye disorders) | 5
Photophobia (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 34
Stomach pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 18
Fatigue (General disorders) | 84
General disorders and administration site conditions - Other (General disorders) | 3
Pain (General disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 46
Fall (Injury, poisoning and procedural complications) | 2
Blood gonadotrophin abnormal (Investigations) | 1
Blood prolactin abnormal (Investigations) | 3
Growth hormone abnormal (Investigations) | 26
Investigations - Other (Investigations) | 1
Weight gain (Investigations) | 9
Weight loss (Investigations) | 4
White blood cell decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 24
Obesity (Metabolism and nutrition disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 1
Growth suppression (Musculoskeletal and connective tissue disorders) | 9
Kyphosis (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 3
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
IVth nerve disorder (Nervous system disorders) | 3
Somnolence (Nervous system disorders) | 2
Abducens nerve disorder (Nervous system disorders) | 2
Ataxia (Nervous system disorders) | 8
Cognitive disturbance (Nervous system disorders) | 28
Concentration impairment (Nervous system disorders) | 10
Dizziness (Nervous system disorders) | 3
Dysarthria (Nervous system disorders) | 1
Dysesthesia (Nervous system disorders) | 1
Dysphasia (Nervous system disorders) | 1
Facial muscle weakness (Nervous system disorders) | 1
Facial nerve disorder (Nervous system disorders) | 2
Headache (Nervous system disorders) | 31
Hydrocephalus (Nervous system disorders) | 1
Hypersomnia (Nervous system disorders) | 1
Intracranial hemorrhage (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 22
Muscle weakness left-sided (Nervous system disorders) | 3
Muscle weakness right-sided (Nervous system disorders) | 2
Nervous system disorders - Other (Nervous system disorders) | 6
Nystagmus (Nervous system disorders) | 5
Oculomotor nerve disorder (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 2
Stroke (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 13
Insomnia (Psychiatric disorders) | 3
Irritability (Psychiatric disorders) | 7
Psychiatric disorders - Other (Psychiatric disorders) | 3
Urinary frequency (Renal and urinary disorders) | 1
Irregular menstruation (Reproductive system and breast disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 75
Dry skin (Skin and subcutaneous tissue disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 9
Hematoma (Vascular disorders) | 1
Vascular disorders - Other (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes